CLINICAL TRIAL: NCT02457897
Title: Thyroid Hormone to Induce Non-Insulin Mediated Glucose Disposal in Patients With Insulin Receptor Mutations
Brief Title: Thyroid Hormone to Induce Non-Insulin Mediated Glucose Disposal in People With Insulin Receptor Mutations
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 150119; 15-DK-0119
Record Dates: First submitted 2015-04-22; First posted 2015-05-29 (Estimated); Results first posted 2019-12-05 (Actual); Last update posted 2019-12-05 (Actual); Status verified 2018-09-18

CONDITIONS: Insulin Resistance; Diabetes Mellitus; Abnormal Glucose Metabolism
Keywords: Brown Adipose Tissue; Liothyronine; Insulin Receptors
MeSH Terms: conditions — Insulin Resistance; Diabetes Mellitus | interventions — Triiodothyronine

ARMS (1):
- Patients with insulin receptor mutation (Experimental)
  Interventions: Drug: Liothyronine

INTERVENTIONS:
Drug: Liothyronine — Oral supplement given every 8 hours

SUMMARY:
Background:

- Insulin receptor mutation causes high blood sugars and sometimes diabetes complications. Researchers want to see if thyroid hormone helps.

Objectives:

- To see if thyroid hormone treatment changes how the body handles sugar in people with insulin receptor mutation and improves blood sugar in people with diabetes.

Eligibility:

- People ages 12 65 with an insulin receptor mutation.

Design:

* Study part 1:19-day clinic stay. Participants will be monitored for 4 days. Then for 15 days they will take a thyroid hormone pill 3 times a day. Participants will have:
* Blood tests.
* Heart rate and skin temperature monitored.
* All their food provided.
* Two 5-hour sessions in a special room. They will wear special clothes and sometimes sit still.
* Two small tubes inserted in veins. One will deliver tiny amounts of sugar and fat with a non-radioactive tracer. Participants will also drink water with a tracer. The other tube will collect blood.
* A sweet drink. Participants may have finger stick blood sugar tests.
* Glucose-monitoring device inserted into body fat for two 24-hour periods.
* Adults may have samples of fat and muscle taken.
* Heart ultrasound.
* PET-CT scan in a machine. An intravenous catheter will be placed in an arm vein. A small amount of radioactive substance will be injected.
* DEXA scan of body fat and bone density.
* Participants with poorly controlled diabetes will then take thyroid hormone at home for 6 months. They will have blood drawn and sent to the study team monthly.
* After about 3 months, they will have an overnight visit. After 6 months, they will have a 4-day visit.

DETAILED DESCRIPTION:
Background

Patients with mutations of the insulin receptor have extreme insulin resistance. This frequently results in diabetes in childhood that is extremely difficult to manage with conventional diabetes therapies, including insulin at doses 10-50 fold higher than usual. Poorly controlled diabetes, in turn, leads to microvascular complications (e.g. blindness) and early death. Hyperthyroidism, whether endogenous (e.g. Graves' disease) or exogenous, increases energy expenditure, activates brown adipose tissue, and enhances skeletal muscle perfusion, leading to enhanced glucose disposal. In a single patient with mutation of the insulin receptor and poorly controlled diabetes despite maximal therapy, iatrogenic mild hyperthyroidism for treatment of thyroid cancer resulted in normalization of glycemic control, suggesting that thyroid hormone treatment could have therapeutic benefit in this rare disease.

Aim

The purpose of this study is to determine if treatment with thyroid hormone will increase glucose disposal in patients with mutations of the insulin receptor, and thereby improve glycemic control. The hypotheses to be tested are:

1. Thyroid hormone will increase whole-body glucose disposal in patients with insulin receptor mutations.
2. This increased glucose disposal will be mediated via increased glucose uptake in brow adipose tissue (BAT) and muscle.
3. Increases in glucose disposal will result in improved glycemic control.

Methods

This study is a non-randomized pre-post design, conducted in two sequential parts. Part 1 is a short-term (2 week) proof-of-principle study to test whether thyroid hormone will increase glucose disposal in patients with insulin receptor mutations (with or without diabetes), and the mechanisms by which increased glucose disposal occurs. Part 2 is a longer term (6 month) therapeutic study to test whether thyroid hormone will result in improved glycemic control in diabetic patients with insulin receptor mutations.

ELIGIBILITY:
* 2 WEEKS STUDY:

INCLUSION CRITERIA:

1. Mutation of the insulin receptor (either recessive or dominant negative). If mutation status is not known prior to enrollment, subjects will undergo genotyping at enrollment. In the unanticipated event that a patient does not have a mutation of the insulin receptor, he or she will not complete the study and his or her data will not be included in the analysis.

EXCLUSION CRITERIA:

1. Changes in doses of diabetes medications (including metformin, insulin, sulfonylureas, thiazolidinediones, leptin, GLP-1 agonists, DPP4 inhibitors, etc.) in the preceding 10 weeks.
2. Any medical condition or medication that will increase risk to the subject (e.g. ischemic or structural heart disease, congestive heart failure, uncontrolled hypertension, or arrhythmia) or that will interfere with interpretation of study data.
3. Disorders that would lead to erratic gastrointestinal absorption or loss of thyroid hormone from the gut (severe diarrhea, celiac disease, use of bile acid sequestrants, excessive consumption of soybean products).
4. Any form of endogenous hyperthyroidism or hypothyroidism at baseline.
5. Current or recent (past 8 weeks) use of thyroid hormone or anti-thyroid drugs.
6. Extreme disorders of thyroid hormone binding to thyroid binding globulin (excess or deficiency) or protein loss (nephrotic range proteinuria) that would lead to difficulties achieving a consistent thyroid hormone level for study.
7. Known presence of a rare clinical disorder that leads to thyroid hormone insensitivity (known T3 receptor mutations, selenocysteine insertion sequence-binding protein 2 (SBP2) abnormalities, monocarboxylate transporter defects).
8. Current use of beta blockers
9. Pregnancy or breast feeding
10. Any EKG abnormality that could increase risk of T3 treatment (resting sinus tachycardia (age adjusted norms), atrial fibrillation, myocardial ischemia, left or right ventricular excitation block, left ventricular hypertrophy or extrasystoles)
11. Known allergy or hypersensitivity to any form of thyroid hormone
12. Known adrenal insufficiency
13. Dependence on oral anticoagulant medications (adults only)
14. Use of tricyclic anti-depressants, as transient cardiac arrhythmias have been observed with the concomitant use of thyroid hormone.
15. Use of cholestyramine.
16. History of clinically significant osteoporosis per investigator judgment (e.g. previous fragility fracture)

6 MONTHS STUDY:

Patients must meet all inclusion and exclusion criteria for the short-term study, plus have poorly controlled diabetes, defined as a hemoglobin A1c greater than or equal to 7%.

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2015-04-17; Primary Completion 2018-09-18 (Actual); Study Completion 2018-09-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca J Brown, M.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Kahn CR, Flier JS, Bar RS, Archer JA, Gorden P, Martin MM, Roth J. The syndromes of insulin resistance and acanthosis nigricans. Insulin-receptor disorders in man. N Engl J Med. 1976 Apr 1;294(14):739-45. doi: 10.1056/NEJM197604012941401. PMID 176581
- [Background] Skarulis MC, Celi FS, Mueller E, Zemskova M, Malek R, Hugendubler L, Cochran C, Solomon J, Chen C, Gorden P. Thyroid hormone induced brown adipose tissue and amelioration of diabetes in a patient with extreme insulin resistance. J Clin Endocrinol Metab. 2010 Jan;95(1):256-62. doi: 10.1210/jc.2009-0543. Epub 2009 Nov 6. PMID 19897683
- [Background] Musso C, Cochran E, Moran SA, Skarulis MC, Oral EA, Taylor S, Gorden P. Clinical course of genetic diseases of the insulin receptor (type A and Rabson-Mendenhall syndromes): a 30-year prospective. Medicine (Baltimore). 2004 Jul;83(4):209-222. doi: 10.1097/01.md.0000133625.73570.54. PMID 15232309
- [Derived] Sekizkardes H, Chung ST, Chacko S, Haymond MW, Startzell M, Walter M, Walter PJ, Lightbourne M, Brown RJ. Free fatty acid processing diverges in human pathologic insulin resistance conditions. J Clin Invest. 2020 Jul 1;130(7):3592-3602. doi: 10.1172/JCI135431. PMID 32191645
- [Derived] Kushchayeva YS, Startzell M, Cochran E, Auh S, Sekizkardes H, Soldin SJ, Kushchayev SV, Dieckmann W, Skarulis M, Abdul Sater Z, Brychta RJ, Cypess AM, Lin TC, Lightbourne M, Millo C, Brown RJ. Thyroid Hormone Effects on Glucose Disposal in Patients With Insulin Receptor Mutations. J Clin Endocrinol Metab. 2020 Mar 1;105(3):e158-71. doi: 10.1210/clinem/dgz079. PMID 31588494
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2015-DK-0119.html

RESULTS

PARTICIPANT FLOW:
Period: Part 1 Short-term (2 Weeks) Study
Arm/Group | Patients With Insulin Receptor Mutation
Started | 7
Completed | 7
Not Completed | 0
Period: Part 2 Long-term (6 Month) Study
Arm/Group | Patients With Insulin Receptor Mutation
Started | 5 (Two patients were not eligible for Part 2 study because their HbA1c was less than 7.)
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Patients With Insulin Receptor Mutation
Number analyzed (Participants) | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 22 (5.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 3
  Black | 2
  White | 2
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 19.84 (8.33)

OUTCOME MEASURES:

1. Primary Outcome: Total Body Glucose Disposal in the Fasting State
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: μmol/kg LBM (Lean Body Mass)/min
Arm/Group | Patients With Insulin Receptor Mutation
Number analyzed (Participants) | 7
μmol/kg LBM (Lean Body Mass)/min | 21.47 (6)

2. Primary Outcome: Hemoglobin A1C
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: percentage of glycosylated hemoglobin
Arm/Group | Patients With Insulin Receptor Mutation
Number analyzed (Participants) | 5
percentage of glycosylated hemoglobin | 9.1 (3)

3. Secondary Outcome: Muscle Glucose Uptake
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: μmol/min/100ml
Arm/Group | Patients With Insulin Receptor Mutation
Number analyzed (Participants) | 5
μmol/min/100ml | 0.9 (0.08)

4. Secondary Outcome: Muscle Glucose Uptake
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: μmol/min/100ml
Arm/Group | Patients With Insulin Receptor Mutation
Number analyzed (Participants) | 2
μmol/min/100ml | 2.0 (0.2)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Patients With Insulin Receptor Mutation
All-Cause Mortality (participants affected / at risk) | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 3/7
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients With Insulin Receptor Mutation (N=7)
Allergic reaction (after eating Indian food) (Immune system disorders) | 1 (1)
Upper Respiratory infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hyperglycemia (Endocrine disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-15): https://cdn.clinicaltrials.gov/large-docs/97/NCT02457897/Prot_SAP_000.pdf